CLINICAL TRIAL: NCT05982431
Title: Kinesiology Taping Helps Patients With First Metatarsophalangeal Joint Sprain
Brief Title: Metatarsophalangeal Joint Sprain Kinesiotaping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0063
Record Dates: First submitted 2023-07-10; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Turf Toe; Metatarsophalangeal (Joint) Sprain
Keywords: turf toe; Metatarsophalangeal Sprain; functional ability; gait parameters; kinesiology taping
MeSH Terms: conditions — Foot Injuries; Sprains and Strains | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exercise group (Experimental): 60-minutes exercise program, three times a week on alternate days for 12 successive weeks.
  Interventions: Other: Traditional physical therapy program
- placebo kinesiology taping plus exercise group (Experimental): Kinesiology taping was used, however the strain was zero. Before each exercise session, the tape was changed every two days while the patients were present.
  Interventions: Other: Traditional physical therapy program; Other: placebo Kinsio taping
- kinesiology taping plus exercise group (Experimental): putting no stress on the opposite end and a 50% stretch from the top of the big toe to the heel along the back of the heel. After applying a 50% stretch from the top of the big toe to the second horizontal little strip between the big toe and second toe, place the ends below the toe diagonally with no stress.
  Interventions: Other: Traditional physical therapy program; Other: Kinsio taping

INTERVENTIONS:
Other: Traditional physical therapy program — 60-minutes exercise program, three times a week on alternate days for 12 successive weeks
  Other Names: exercise program
Other: Kinsio taping — One full strip of kinesiology taping tape and one half-length strip were needed for the kinesiology taping application
  Other Names: kinesiology taping
  Arms: kinesiology taping plus exercise group
Other: placebo Kinsio taping — One full strip of kinesiology taping tape and one half-length strip were needed for the placebo kinesiology taping application
  Other Names: placebo kinesiology taping
  Arms: placebo kinesiology taping plus exercise group

SUMMARY:
kinesio taping would reduce pain, improve gait performance, and enhance the functional capacity of turf toe patients undergoing physical therapy

DETAILED DESCRIPTION:
Health practitioners have recently become interested in using kinesiology taping in clinical practice as an alternative to traditional taping and bracing procedures for treating a variety of diseases, including sprain of metatarsophalangeal joint of the big toe. Patients with turf toe can benefit from kinesiology tape because it offers therapeutic support and stability while preserving a normal range of motion.

ELIGIBILITY:
Inclusion Criteria:

* comprised athletes with 2nd grade turf toe.
* medically stable.
* had foot pain for more than a month prior to enrollment.
* didn't have persistent, incapacitating pain.
* had a doctor's note approving their decision to stop taking painkillers during the research.

Exclusion Criteria:

* if they had any surgical intervention before.
* range of motion limitation in the ankle joint.
* inability to exercise.
* systemic disease.
* any other orthopedic problem at ankle joints.

Ages: 25 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Pain visual analog scale | at first week
  The degree of the pain was assessed using a 10-cm visual analog scale (VAS), with 0 denoting no pain and 10 denoting the most painful event.
Pain visual analog scale | after 12 weeks
  The degree of the pain was assessed using a 10-cm visual analog scale (VAS), with 0 denoting no pain and 10 denoting the most painful event.
Gait parameters (step length by centimeter). | at first week
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.
Gait parameters (step length by centimeter). | after 12 weeks
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.
Gait parameters (stride length by meter). | at first week
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.
Gait parameters (stride length by meter). | after 12 weeks
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.
Gait parameters (cadence by steps per minute). | at first week
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.
Gait parameters (cadence by steps per minute). | after 12 weeks
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.
Gait parameters (velocity by centimeter per second). | at first week
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.
Gait parameters (velocity by centimeter per second). | after 12 weeks
  The twelve computerized cameras of the VICON 3D motion analysis system were used to record gait data.

SECONDARY OUTCOMES:
Functional ability assessment | at first week
  Functional ability was assessed using the 6-minute walk test.
Functional ability assessment | after 12 weeks
  Functional ability was assessed using the 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa Azab, PhD, Principal Investigator — Cairo University
Locations (2):
- Saudi Arabia (2):
  - Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region
  - King Khalid Hospital, Al Kharj, Riyadh Region

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Mostafavifar M, Wertz J, Borchers J. A systematic review of the effectiveness of kinesio taping for musculoskeletal injury. Phys Sportsmed. 2012 Nov;40(4):33-40. doi: 10.3810/psm.2012.11.1986. PMID 23306413
- [Background] Burr JF, Bredin SS, Faktor MD, Warburton DE. The 6-minute walk test as a predictor of objectively measured aerobic fitness in healthy working-aged adults. Phys Sportsmed. 2011 May;39(2):133-9. doi: 10.3810/psm.2011.05.1904. PMID 21673494
- [Background] Kim MK, Shin YJ. Immediate Effects of Ankle Balance Taping with Kinesiology Tape for Amateur Soccer Players with Lateral Ankle Sprain: A Randomized Cross-Over Design. Med Sci Monit. 2017 Nov 21;23:5534-5541. doi: 10.12659/msm.905385. PMID 29158472